CLINICAL TRIAL: NCT00659230
Title: A Randomized, Placebo-Controlled Trial of the Dopamine-B-Hydroxylase (DBH) Inhibitor, Nepicastat, for the Treatment of PTSD in OIF/OEF Veterans
Brief Title: Nepicastat for Posttraumatic Stress Disorder (PTSD) in OIF/OEF Veterans
Acronym: Nepicastat
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tuscaloosa Research & Education Advancement Corporation (Other)
Collaborators: Acorda Therapeutics (Industry); Ralph H. Johnson VA Medical Center (U.S. Federal Agency); Baylor College of Medicine (Other); San Diego Veterans Healthcare System (U.S. Federal Agency); James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lori Davis, MD, Associate Chief of Staff, Tuscaloosa Research & Education Advancement Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-06; PT074384/W81XWH-08-2-0071 (Other Grant/Funding Number: Department of Defense/USAMRAA); PT074384/W81XWH-09-1-0287 (Other Grant/Funding Number: Department of Defense/USAMRAA)
Record Dates: First submitted 2008-03-10; First posted 2008-04-16 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-09

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Veterans; Nepicastat; OIF/OEF
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — nepicastat; Dopamine beta-Hydroxylase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Arm 1
  Interventions: Drug: Placebo
- Nepicastat (Active Comparator): Arm 2
  Interventions: Drug: Nepicastat

INTERVENTIONS:
Drug: Nepicastat — 100-800mg
  Other Names: SYN117; Dopamine beta hydroxylase (DBH) inhibitor
  Arms: Nepicastat
Drug: Placebo — 100-800mg placebo
  Arms: Placebo

SUMMARY:
This study proposes a multi-site, randomized, double-blind, placebo-controlled clinical trial of the dopamine-ß-hydroxylase (DBH) inhibitor, nepicastat, for the treatment of posttraumatic stress disorder (PTSD) in outpatients who have previously served in a combat zone during Operation Iraqi Freedom and Operation Enduring Freedom (OIF/OEF)or other Southwest conditions since 19800. A DBH inhibitor's mechanism of action is to decrease neuronal noradrenaline (NA) release by inhibiting DBH conversion of dopamine (DA) to NA. Animal models of PTSD and human studies have found a substantial increase in NA activity for these animal models and for PTSD in humans. Furthermore, recent clinical studies have improved PTSD hyper-arousal symptoms by reducing the NA over-activity using agents like NA post-synaptic antagonists. Key support for the proposed study is based on a similar improvement in PTSD symptoms after treatment with the DBH inhibitor, disulfiram.

In the experience of the clinical investigators, the most common chief complaint of the OIF/OEF veterans with PTSD is hyperarousal (DSM-IV criterion D symptom cluster). These symptoms significantly interfere with social, occupational, and interpersonal function. Standard treatments with antidepressants are not fully effective in treating the symptoms of PTSD in veterans; thus, new treatments are needed. An intervention, such as nepicastat, aimed at reducing hyperarousal, as well as other PTSD symptoms, would have significant impact of restoring overall function and quality of life in OIF/OEF veterans with PTSD. Since hyperarousal symptoms responded relatively quickly to medications of this type, our study in 120 outpatient veterans with PTSD will compare nepicastat 120 mg/day vs. placebo in a 6-week double-blind, randomized clinical trial (RCT). The veterans will be followed for an additional 8 weeks after the RCT, during which, those who have a priori defined positive clinical response to the study medication, nepicastat vs. placebo, will be continued on the study medication, in order to assess further improvement and safety. Those patients who do not have a positive clinical response during the 6 week RCT will be offered the addition of the standard first-line PTSD pharmacotherapy, paroxetine, during the 8 weeks extension phase. Thus, weeks 7-14 offer an opportunity to evaluate longer-term nepicastat efficacy and to compare the treatment response of nonresponders after augmentation with paroxetine.

DETAILED DESCRIPTION:
HYPOTHESES Primary Hypothesis: Compared to placebo treatment, nepicastat-treated OIF/OEF veterans with PTSD will have significantly reduced PTSD hyperarousal symptoms as defined by the Clinician Administered PTSD Scale [CAPS], subscale D (CAPS-D).

Secondary Hypotheses: Compared to placebo, nepicastat-treated OIF/OEF veterans with PTSD will have:

* Significantly reduced PTSD symptoms (total CAPS)
* Significantly reduced PTSD reexperiencing symptoms (CAPS-B)
* Significantly reduced PTSD avoidance symptoms (CAPS-C)

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patient understands the risks and benefits and agrees to visit frequency and procedures
* Male or female
* Any race or ethnic origin
* Served in OIF/OEF or Afghanistan conflicts or other Southwest Asia conditions
* Currently Active Duty, National Guard, Reservist, Veteran, and/or Retired Military
* Diagnosis of PTSD (by MINI (Mini International Neuropsychiatric Interview) and CAPS-DX (Clinician Administered PTSD scale- Diagnostic Form) using Rule of Fours and total CAPS-DX score of 45)
* No substance use disorders in the previous 2 weeks and no substance dependence disorders in the past 4 weeks (except for nicotine and caffeine)
* Free of psychotropic medication for 2 weeks prior to randomization
* Physical and laboratory panel are within normal limits or not clinically significant
* Women of childbearing potential must be using medically-approved methods of birth control
* ≥19 to 65 years of age

Exclusion Criteria:

* Lifetime history of bipolar I, schizophrenia, schizoaffective or cognitive disorders
* Actively considering plans of suicide or homicide
* Psychotic symptoms that in the investigator's opinion impair the patient's ability to give informed consent or make it unsafe for patient to be maintained without a neuroleptic
* Unstable general medical conditions or a contraindication to the use of nepicastat
* Women planning to become pregnant or breastfeed during the study
* Current or pending incarceration
* Terminal Illness

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2012-07-05 (Actual); Study Completion 2012-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Berry, M.D., Study Chair — IRB Tuscaloosa VAMC
Locations (3):
- United States (3):
  - Tuscaloosa VAMC, Tuscaloosa, Alabama
  - VA San Diego Healthcare System, San Diego, California
  - James J.Peters VA Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kosten TR, Krystal J. Biological mechanisms in posttraumatic stress disorder. Relevance for substance abuse. Recent Dev Alcohol. 1988;6:49-68. doi: 10.1007/978-1-4615-7718-8_3. PMID 3283864
- [Background] Graham DP, Nielsen DA, Kosten TR, Davis LL, Hamner MB, Makotkine I, Yehuda R. Examining the utility of using genotype and functional biology in a clinical pharmacology trial: pilot testing dopamine beta-hydroxylase, norepinephrine, and post-traumatic stress disorder. Psychiatr Genet. 2014 Aug;24(4):181-2. doi: 10.1097/YPG.0000000000000039. No abstract available. PMID 24983834

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Nepicastat
Started | 51 (2 did not return post-randomization, 5 lost source documents, thus 7 excluded from results analysis) | 49 (3 did not return post-randomization, 4 lost source documents, thus 7 excluded from results analysis)
Completed | 42 | 37
Not Completed | 9 | 12
Not completed — Lost to Follow-up | 2 | 5
Not completed — Lost source documentation | 5 | 4
Not completed — Did not return post-randomization | 2 | 3

BASELINE CHARACTERISTICS:
Population: Placebo: 2 did not return post-randomization & were excluded from outcome analysis; 5 lost source documents & were excluded from baseline, safety, & outcomes analyses. Nepicastast: 3 did not return post-randomization and were excluded from outcome analysis, 4 lost source documents and were excluded from baseline, safety, and outcome analyses
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nepicastat | Total
Number analyzed (Participants) | 46 | 45 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.61 (10.49) | 39.33 (11.01) | 37.96 (10.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 42 | 44 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 44 | 40 | 84
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 22 | 44
  White | 21 | 16 | 37
  More than one race | 3 | 7 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 46 | 45 | 91
CAPS-D Score (primary outcome) [Mean (Standard Deviation); unit: units on a scale] — CAPS-D is the subscore for the hyperarousal symptoms cluster of PTSD; higher score is more severe; range is 0-40.
  units on a scale | 25.59 (6.17) | 26.07 (6.01) | 25.82 (6.06)

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale Subscore D (Hyperarousal)
Description: The Clinician Administered PTSD Scale subscore D (CAPS-D) measures the hyperarousal cluster for PTSD symptoms (5 items). Higher scores indicate greater severity. Range for CAPS-D is zero to 40. The CAPS has acceptable test-retest reliability (0.98), sensitivity (0.84), specificity (0.95), internal consistency (0.76-0.88) and validity (κ=0.78).
Time Frame: Baseline, week 2, 4 and 6
Population: Participants who returned for at least one post-randomization visit and had source documentation (in placebo group 2 did not return and the source documentation for 5 participants was lost; for nepicastat group 3 did not return and the source documentation for 4 participants was lost).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Nepicastat
Number analyzed (Participants) | 44 | 42
units on a scale
  Baseline | 25.59 (6.17) | 26.07 (6.01)
  Week 2 | 21.20 (7.59) | 22.07 (7.95)
  Week 4 | 19.78 (8.27) | 21.15 (8.13)
  Week 6 | 19.57 (8.55) | 21.62 (9.17)
Statistical Analysis 1: Comparison: Placebo vs Nepicastat; The analysis was conducted using a repeated-measures analysis of variance (ANOVA) model. The model consisted of two factors - treatment at two levels and time (5 time points including baseline) and group by time interaction; Test type: Superiority or Other; p = 0.723, ANOVA; Effect Size = -0.18, 90% CI 2-sided [-0.64 to 0.27] — Effect size (ES) for change in CAPS-D score relative to baseline was calculated according to the method of Cohen

2. Secondary Outcome: Clinician Administered PTSD Scale Total Score
Description: The Clinician Administered PTSD Scale (CAPS) measures the full spectrum of PTSD symptoms. Higher scores indicate greater severity. Range for CAPS is zero to 136. The CAPS has acceptable test-retest reliability (0.98), sensitivity (0.84), specificity (0.95), internal consistency (0.76-0.88) and validity (κ=0.78).
Time Frame: Baseline, week 2,4, and 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Nepicastat
Number analyzed (Participants) | 44 | 42
units on a scale
  Baseline | 74.52 (16.73) | 77.18 (16.55)
  Week 2 | 61.82 (25.02) | 60.17 (24.72)
  Week 4 | 52.61 (27.17) | 60.26 (27.59)
  Week 6 | 58.22 (28.37) | 52.95 (25.81)
Statistical Analysis 1: Comparison: Placebo vs Nepicastat; Test type: Superiority; p = 0.540, ANOVA; Effect Size = -0.07, 90% CI 2-sided [-.52 to 0.39] — Effect size (ES) for change in CAPS-D score relative to baseline was calculated according to the method of Cohen

3. Secondary Outcome: Clinician Administered PTSD Scale Subscale B Score
Description: The Clinician Administered PTSD Subscale B (CAPS-B) measures the re-experiencing cluster of PTSD symptoms. Higher scores indicate greater severity. Range for CAPS-B is zero to 40. The CAPS has acceptable test-retest reliability (0.98), sensitivity (0.84), specificity (0.95), internal consistency (0.76-0.88) and validity (κ=0.78). Blake, D.D., Weathers, F.W., Nagy, L.M., Kaloupek, D.G., Gusman, F.D., Charney, D.S., Kean, T.M., 1995, The development of a clinician-administered PTSD scale. Journal of Traumatic Stress, 8:75-90.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Nepicastat
Number analyzed (Participants) | 44 | 42
units on a scale
  Baseline | 20.37 (7.26) | 20.41 (8.46)
  Week 2 | 16.95 (9.77) | 14.14 (8.97)
  Week 4 | 11.51 (10.02) | 14.59 (9.75)
  Week 6 | 12.64 (10.04) | 15.27 (10.27)
Statistical Analysis 1: Comparison: Placebo vs Nepicastat; Test type: Superiority; p = 0.951, ANOVA; Effect size = -0.18, 90% CI 2-sided [-0.64 to 0.27] — Effect size (ES) for change in CAPS-D score relative to baseline was calculated according to the method of Cohen

4. Secondary Outcome: Clinician Administered PTSD Scale Subscale C Score
Description: The Clinician Administered PTSD Subscale C (CAPS-C) measures the Avoidance and emotional numbing cluster of PTSD symptoms. Higher scores indicate greater severity. Range for CAPS-C is zero to 56. The CAPS has acceptable test-retest reliability (0.98), sensitivity (0.84), specificity (0.95), internal consistency (0.76-0.88) and validity (κ=0.78).
Time Frame: Baseline, week 2, 4, and 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Nepicastat
Number analyzed (Participants) | 44 | 42
units on a scale
  Baseline | 29.02 (8.03) | 30.70 (7.37)
  Week 2 | 23.66 (12.18) | 24.39 (11.41)
  Week 4 | 21.32 (12.82) | 24.51 (13.06)
  Week 6 | 20.74 (12.21) | 21.32 (12.11)
Statistical Analysis 1: Comparison: Placebo vs Nepicastat; Test type: Superiority; p = 0.396, ANOVA; Effect Size = 0.11, 90% CI 2-sided [-0.35 to 0.56] — Effect size (ES) for change in CAPS-D score relative to baseline was calculated according to the method of Cohen

ADVERSE EVENTS:
Time Frame: During six-week placebo-controlled phase.
Description: Adverse events were defined the same as clinicaltrials.gov. Adverse events were systematically assessed at each research visit for type of adverse event, length of time, severity, action taken, and relatedness to study medication. The source documentation was lost for 9 participants at one site (5 placebo and 4 nepicastat) and were not included in safety analysis.
Arm/Group | Placebo | Nepicastat
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/45
Serious Adverse Events (participants affected / at risk) | 3/46 | 2/45
Other Adverse Events (participants affected / at risk) | 25/46 | 27/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=46) | Nepicastat (N=45)
Chest Pain (Cardiac disorders) | 1 (2) | 1 (1) — Hospitalized for Chest Pain
Psychiatric Inpatient (Psychiatric disorders) | 2 (2) | 1 (1) — Mental Illness; Substance Use
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=46) | Nepicastat (N=45)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 7 (7)
Dry Eye (Eye disorders) | 0 (0) | 1 (1)
Gastroesophageal Reflux (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomitting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 3 (3) | 0 (0)
Edema Face (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Flu-like (Infections and infestations) | 5 (5) | 4 (5)
sinusitis (Infections and infestations) | 1 (1) | 2 (2)
MRSA staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
injury to extremity (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
muscle twitch (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
headache (Nervous system disorders) | 7 (7) | 9 (9)
dysgeusia (taste changes) (Nervous system disorders) | 1 (1) | 0 (0)
paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
memory problems (Nervous system disorders) | 0 (0) | 1 (1)
insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
tongue lesion removed (Surgical and medical procedures) | 1 (1) | 0 (0)
superficial thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 0 (0) | 1 (1)
hot flash (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations: short duration of placebo-controlled phase (six-weeks).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No